CLINICAL TRIAL: NCT06156566
Title: European Randomised Clinical Trial on mPOX Infection
Brief Title: European Trial Into Mpox Infection
Acronym: EPOXI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Miquel Ekkelenkamp (Other)
Collaborators: European Clinical Research Alliance for Infectious Diseases (ECRAID) (Other); Erasmus Medical Center (Other); Hospital Universitario La Paz (Other); ANRS, Emerging Infectious Diseases (Other Government); Universiteit Antwerpen (Other)
Responsible Party: Sponsor-Investigator, Miquel Ekkelenkamp, Clinical Microbiologist, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-501979-10
Record Dates: First submitted 2023-10-25; First posted 2023-12-05 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-08

CONDITIONS: Monkeypox
Keywords: tecovirimat; mpox; TPOXX
MeSH Terms: conditions — Mpox, Monkeypox | interventions — tecovirimat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial is controlled with matching placebo. Unblinding after database lock.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tecovirimat (Active Comparator): Oral treatment with tecovirimat 200 mg capsules. Twice daily three capsules orally. Duration of treatment: 14 days (28 administrations).
  Interventions: Drug: Tecovirimat Oral Capsule
- Placebo (Placebo Comparator): Matching placebo to tecovirimat capsules. Twice daily three capsules orally. Duration of treatment: 14 days (28 administrations).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tecovirimat Oral Capsule — 600 mg, twice daily, 14 days.
  Other Names: Tpoxx Tecovirimat
  Arms: Tecovirimat
Drug: Placebo — 3 capsules, twice daily, 14 days.
  Other Names: Oral placebo capsule
  Arms: Placebo

SUMMARY:
The goal of this randomized controlled double-blind clinical trial is to test the drug tecovirimat in patients with mpox (previously known as monkeypox) disease.

The main questions it aims to answer are:

* Is tecovirimat effective in treating mpox infection.
* Is tecovirimat safe to treat patients with mpox infection.

Participants will receive either the drug tecovirimat orally, 600 mg twice per day, or a matching placebo. The outcome of the infection and the side effect experienced will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Polymerase Chain Reaction (PCR) /Nucleic Acid Amplification Test (NAAT) -confirmed mpox infection
* The presence of active skin or mucosal lesion(s)
* Signed Informed Consent Form

Exclusion Criteria:

* Age <18 years.
* Body weight <40 kg
* Pregnant and breastfeeding patients are not eligible for inclusion in this study.
* Lack of mental capacity to provide informed consent
* Trial participation is considered not in the best interest of patient
* Known hypersensitivity to the active substance or to any of the excipients of the study drug.
* Use of contraindicated treatment repaglinide. (Repaglinide, an oral treatment for diabetes mellitus, may be discontinued while taking study treatment with the agreement of the patient's general practitioner, who may start alternate diabetes treatment if considered necessary.)
* Previous, current or planned use of another investigational drug (tecovirimat) at any point during study participation.
* The patient's own doctor considers there to be a definite indication for the patient to receive tecovirimat or the local guidelines establish that tecovirimat treatment should be initiated
* The patient's own doctor considers there to be a definite contraindication to the patient receiving tecovirimat.
* The patient suffers from hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Time to complete mpox lesion resolution | 28 days
  Time in days until day 28 after randomization, until the first day on which all lesions are completely healed with a new fresh layer of skin.

SECONDARY OUTCOMES:
Time to active lesion resolution | 28 days
  The first day on which all skin lesions are scabbed or desquamated (and mucosal lesions healed), counted from start of therapy, with follow-up up to 28 days after randomisation
Status of the lesions on day 7, 14 and 28 | Day 7, day 14 and day 28
  Status of the lesions on day 7, 14, 21 and 28 according to an ordinal scale. The ordinal scale is a) all lesions completely resolved (all scabs dropped off and intact skin remains underneath, and all mucosal lesions healed), b) active lesions resolved (all skin lesions scabbed or desquamated, but not fully resolved), c) active lesions persist but no new lesions in last 24 hours, d) new lesion(s) in last 24 hours.
Time to resolution of symptoms | 90 days
  Time to resolution of symptoms. Symptoms are counted from start of therapy and assessed by self-assessment. These include fatigue, malaise, nausea, vomiting, abdominal pain, anorexia, cough, dysphagia, odynophagia, fever, headache, oral pain, pain with urination, rectal/anal pain. Signs will be evaluated at study visits only, including lymphadenopathy and proctitis, and are not included in the evaluation of symptoms.
Occurrence of a negative monkeypox PCR of skin or mucosal swab | Days 7, 14 and 28
  Negative monkeypox PCR (Polymerase Chain Reaction) of skin or mucosal swab, assessed for the two most active skin lesions or for the mucosal lesion.
Persistence of scars and skin discoloration | Assessed on day 90
  Assessment of scars and/or skin discoloration of mpox lesions.
Change from baseline in quality of life | Assessed on day 14 and day 90.
  Change from baseline of quality of life, assessed by the Dermatology Life Quality Index (DLQI).
  Minimum value = 0, maximum value = 30, a higher score indicates a worse outcome. (Ten questions with each a minimum of 0 and a maximum of 3.)
All-cause mortality | Assessed on day 28 and on day 90
  All-cause mortality
Time to complication or all-cause admission to hospital or all-cause death | Assessed within 28 days and within 90 days.
  Time to complication or all-cause admission to hospital or all-cause death, within 28 days and within 90 days, applicable to outpatients only, and counted from start of therapy. A complication includes genitourinary complications (e.g. urinary retention, paraphimosis), lower respiratory tract complication (e.g. pneumonia and need for oxygen), ocular impairment (e.g. keratitis), neurologic impairment (e.g. encephalitis) or mental health disturbance (e.g. confusion), cardiac impairment (e.g. cardiomyopathy or myocarditis), severe dehydration needing admission, secondary bacterial skin infection or severe pain needing hospital admission.
Frequency of AEs, SAEs and SUSARs | Assessed within 28 days and within 90 days.
  Frequency of Adverse Events (AEs), Serious Adverse Events (SAEs) and Suspected Unexpected Serious Adverse Reaction (SUSARs) for the specific therapeutic, within the first 28 days, but also assessed during the total follow-up (up to day 90).
Resolution of pain | Assessed on days 7, 14 and 90.
  Resolution of pain, by measuring:
  1. time to resolution of pain assessed by the Numeric Rating Scale (NRS) for pain,
  2. time to cessation of the use of analgesic medication, defined as time to consistently reporting no use of analgesia for mpox-related lesions, up to 90 days after randomisation.
  3. anal pain on days 7, 14, and 90 assessed by the Health Related Symptom Index.

CONTACTS AND LOCATIONS:
Overall Officials: Miquel B Ekkelenkamp, MD, PhD, Principal Investigator — UMC Utrecht
Locations (12):
- Belgium (2):
  - Institute of Tropical Medicine, Antwerp, Antwerp
  - Cliniques Universitaires St. Luc, Brussels
- APHP St. Louis, Paris, France
- Universitätsklinikum Bonn, Bonn, Germany
- Italy (2):
  - Hospital Luigi Sacco, Milan
  - Azienda Ospedaliera Universitaria Integrata Verona - AOUI Verona, Verona
- Amsterdam UMC - AMC, Amsterdam, Netherlands
- Oslo Unversity Hospital, Oslo, Norway
- Hospital de Santo António dos Capuchos, Lisbon, Portugal
- Spain (3):
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen Macarena, Seville

REFERENCES:
- [Background] Wedekind C. The infectivity, growth, and virulence of the cestode Schistocephalus solidus in its first intermediate host, the copepod Macrocyclops albidus. Parasitology. 1997 Sep;115 ( Pt 3):317-24. doi: 10.1017/s0031182097001406. PMID 9300470
- [Background] Jang TJ, Lee JI, Kim JR, Kim DH, Bae SH. Decreased gastric proliferation of foveolar epithelial cells after the eradication of Helicobacter pylori. J Korean Med Sci. 1997 Oct;12(5):421-6. doi: 10.3346/jkms.1997.12.5.421. PMID 9364300
- [Background] Benjamini Y, Hochberg Y. Controlling the false discovery rate: a practical and powerful approach to multiple testing. J R Statist Soc B 1995;57(1):289-300.
- [Background] Horton JA, Cruess DF, Romans MC. Compliance with mammography screening guidelines: 1995 Mammography Attitudes and Usage Study Report. Womens Health Issues. 1996 Sep-Oct;6(5):239-45. doi: 10.1016/1049-3867(96)00037-0. No abstract available. PMID 8870502
- [Background] Zherbin EA, Chukhlovin AB. [Loss of specific membrane receptors during the interphase death of thymus cells]. Tsitologiia. 1984 Aug;26(8):973-7. Russian. PMID 6093301
- [Background] Asaki S, Hatori S, Iwai S, Nishimura T, Sato A, Goto Y. Diagnosis of submucosal tumors by injecting a water soluble contrast medium: basic research and imaging of tumors. Tohoku J Exp Med. 1982 Oct;138(2):121-30. doi: 10.1620/tjem.138.121. PMID 7179270
- [Background] EMA: An overview of Tecovirimat SIGA and why it is authorised in the EU. 31-May-2022: https://www.ema.europa.eu/en/documents/overview/tecovirimat-siga-epar-medicine-overview_en.pdf
- [Background] EMA: Summary of product characteristics: www.ema.europa.eu/en/documents/product-information/tecovirimat-siga-epar-product-information_en.pdf, accessed 6-9-2022
- [Background] Mock M, Miyada CG, Collier RJ. Genetic analysis of the functional relationship between colicin E3 and its immunity protein. J Bacteriol. 1984 Aug;159(2):658-62. doi: 10.1128/jb.159.2.658-662.1984. PMID 6086581
- [Background] Grohmann M, Henseling M. Lack of differences between the neuronal and extraneuronal handling of 3H-7- and 3H-ring-2,5,6-(-)noradrenaline. Naunyn Schmiedebergs Arch Pharmacol. 1988 Aug;338(2):180-4. doi: 10.1007/BF00174867. PMID 3185746
- [Background] Hoy SM. Tecovirimat: First Global Approval. Drugs. 2018 Sep;78(13):1377-1382. doi: 10.1007/s40265-018-0967-6. PMID 30120738
- [Background] Howard G, Waller JL, Voeks JH, Howard VJ, Jauch EC, Lees KR, Nichols FT, Rahlfs VW, Hess DC. A simple, assumption-free, and clinically interpretable approach for analysis of modified Rankin outcomes. Stroke. 2012 Mar;43(3):664-9. doi: 10.1161/STROKEAHA.111.632935. Epub 2012 Feb 16. PMID 22343650
- [Background] Jezek Z, Nakano JH, Arita I, Mutombo M, Szczeniowski M, Dunn C. Serological survey for human monkeypox infections in a selected population in Zaire. J Trop Med Hyg. 1987 Feb;90(1):31-8. PMID 3029395
- [Background] Joint ECDC-WHO Regional Office for Europe Monkeypox Surveillance Bulletin, published 31-8-2022: monkeypoxreport.ecdc.europa.eu, accessed 6-9-2022
- [Background] Tritrakarn A. Pulmonary sequestration: ultrasonographic visualization of feeding artery. J Med Assoc Thai. 1989 Aug;72(8):465-8. PMID 2681496
- [Background] Mitchell DL. The induction and repair of lesions produced by the photolysis of (6-4) photoproducts in normal and UV-hypersensitive human cells. Mutat Res. 1988 Nov;194(3):227-37. doi: 10.1016/0167-8817(88)90024-7. PMID 3185582
- [Background] Karcioglu O, Topacoglu H, Dikme O, Dikme O. A systematic review of the pain scales in adults: Which to use? Am J Emerg Med. 2018 Apr;36(4):707-714. doi: 10.1016/j.ajem.2018.01.008. Epub 2018 Jan 6. PMID 29321111
- [Background] Label FDA: https://www.accessdata.fda.gov/drugsatfda_docs/label/2022/214518s000lbl.pdf, accessed 6-9-2022
- [Background] McCullagh P. Regression models for ordinal data (with discussion). J R Statist Soc B. 1980;42:109-42.
- [Background] Germer A, Jahnke C, Mack A, Enzmann V, Reichenbach A. Modification of glutamine synthetase expression by mammalian Muller (glial) cells in retinal organ cultures. Neuroreport. 1997 Sep 29;8(14):3067-72. doi: 10.1097/00001756-199709290-00012. PMID 9331915
- [Background] Wienberg J, Stanyon R, Nash WG, O'Brien PC, Yang F, O'Brien SJ, Ferguson-Smith MA. Conservation of human vs. feline genome organization revealed by reciprocal chromosome painting. Cytogenet Cell Genet. 1997;77(3-4):211-7. doi: 10.1159/000134579. PMID 9284919
- [Background] Pittman PR, Martin JW, Kingebeni PM, Tamfum J-JM, Wan Q, Reynolds MG, et al. Clinical characterization of human monkeypox infections in the Democratic Republic of the Congo. medRxiv. 2022:2022.05.26.22273379.
- [Background] Product Development Under the Animal Rule - Guidance for Industry, FDA October 2015: https://www.fda.gov/media/88625/download, accessed 6-9-2022
- [Background] Kuznetsov VG. [Contamination of vegetables and the external environment of vegetable store houses of the Primor'e Territory by Yersinia]. Gig Sanit. 1986 May;(5):69-71. No abstract available. Russian. PMID 2941342
- [Background] Sale TA, Melski JW, Stratman EJ. Monkeypox: an epidemiologic and clinical comparison of African and US disease. J Am Acad Dermatol. 2006 Sep;55(3):478-81. doi: 10.1016/j.jaad.2006.05.061. PMID 16908354
- [Background] Siegrist EA, Sassine J. Antivirals With Activity Against Mpox: A Clinically Oriented Review. Clin Infect Dis. 2023 Jan 6;76(1):155-164. doi: 10.1093/cid/ciac622. PMID 35904001
- [Background] Cushing M. Who's responsible for too-early discharge? Am J Nurs. 1989 Apr;89(4):471-2. No abstract available. PMID 2650551
- [Background] Tarin-Vicente EJ, Alemany A, Agud-Dios M, Ubals M, Suner C, Anton A, Arando M, Arroyo-Andres J, Calderon-Lozano L, Casan C, Cabrera JM, Coll P, Descalzo V, Folgueira MD, Garcia-Perez JN, Gil-Cruz E, Gonzalez-Rodriguez B, Gutierrez-Collar C, Hernandez-Rodriguez A, Lopez-Roa P, de Los Angeles Melendez M, Montero-Menarguez J, Munoz-Gallego I, Palencia-Perez SI, Paredes R, Perez-Rivilla A, Pinana M, Prat N, Ramirez A, Rivero A, Rubio-Muniz CA, Vall M, Acosta-Velasquez KS, Wang A, Galvan-Casas C, Marks M, Ortiz-Romero PL, Mitja O. Clinical presentation and virological assessment of confirmed human monkeypox virus cases in Spain: a prospective observational cohort study. Lancet. 2022 Aug 27;400(10353):661-669. doi: 10.1016/S0140-6736(22)01436-2. Epub 2022 Aug 8. PMID 35952705
- [Background] Thornhill JP, Barkati S, Walmsley S, Rockstroh J, Antinori A, Harrison LB, Palich R, Nori A, Reeves I, Habibi MS, Apea V, Boesecke C, Vandekerckhove L, Yakubovsky M, Sendagorta E, Blanco JL, Florence E, Moschese D, Maltez FM, Goorhuis A, Pourcher V, Migaud P, Noe S, Pintado C, Maggi F, Hansen AE, Hoffmann C, Lezama JI, Mussini C, Cattelan A, Makofane K, Tan D, Nozza S, Nemeth J, Klein MB, Orkin CM; SHARE-net Clinical Group. Monkeypox Virus Infection in Humans across 16 Countries - April-June 2022. N Engl J Med. 2022 Aug 25;387(8):679-691. doi: 10.1056/NEJMoa2207323. Epub 2022 Jul 21. PMID 35866746
- [Background] WHO fact sheet: www.who.int/news-room/fact-sheets/detail/monkeypox, accessed 6-9-2022
- [Background] I.G. stimulants of the central nervous system. Behav Neuropsychiatry. 1975 Apr-1976 Mar;7(1-12):79-80. No abstract available. PMID 1235851